CLINICAL TRIAL: NCT06046599
Title: Remote Home Assessment of Patients With Amyotrophic Lateral Sclerosis
Acronym: RHAALS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Imperial College London (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 296187
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients living with amyotrophic lateral sclerosis: Individuals with a known diagnosis of amyotrophic lateral sclerosis will be recruited from King's College Hospital's Motor Nerve Clinic. The cohort will contain 20 individuals and their study partners and will be part of the study for one year.

SUMMARY:
The goal of this observational study is the develop new ways of remotely monitoring the health and symptoms of people living with amyotrophic lateral sclerosis from within their homes. The main questions it aims to answer are:

* Can we integrate a new muscle monitoring device into Imperial College London's home monitoring platform?
* Can we investigate and understand the relationship between muscle activity and measure of patient behaviour (e.g., patient movement), physiology (e.g., pulse/blood pressure variation) and sleep quality from the home?
* Can we establish a home-based multimodal biomarker that tracks the neurodegenerative process in ALS? Participants will have passive internet-of-things sensors and internet-enabled medical devices installed in their homes for one year. Some sensors will record automatically without any interaction from the participants, but some will require participants to engage with daily (e.g., blood pressure monitor) on their own or with the help of a study partner.

Where possible, researchers will compare the collected data to other neurodegenerative diseases and healthy controls to understand differences over time.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS), is a neurodegenerative disease that affects nerve cells causing loss of muscle control. Patients with ALS often die within three years of diagnosis. There is only one available drug for ALS, which offers only a small increase to survival by two to three months. The discovery of new drugs for ALS is difficult due to a lack of objective measures that can be used to track disease progression. Consequently, there is a huge need to discover measures that can reliably track ALS over time, which can then be included in clinical trials to speed up drug discovery.

Muscle twitches are a distinctive characteristic present in all patients with ALS. These muscle twitches can be seen at the surface of the skin and can be detected accurately with electromyography (EMGs). We predict that these muscle twitches will provide a sensitive measure of disease progression.

Due to large dropout rates caused by travelling to and from the hospital, we have built and validated a compact high-density EMG device that sits on the surface of the skin to facilitate repeated assessments from patients' homes. This small device is a tenth of the cost of current devices and has been demonstrated to safely and effectively record muscle twitches. The EMG will be integrated into a digital remote home monitoring platform called Minder. Minder is an established platform for recording internet-enabled medical devices and sensors from within a patient's home.

This study aims to establish a home-based digital measure that can track disease progression in patients with ALS. We will recruit 20 patients with ALS from King's Motor Nerve Clinic. Patients will participate in the study for 12-months and will undergo continuous monitoring through the digital monitoring platform alongside regular EMG recordings.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or above at the time of signing the informed consent.
* Diagnosed with ALS by a neurologist with expertise in ALS (Brooks et al., 2000). For subjects with bulbar onset there must be objective limb involvement of at least one limb.
* Diagnosed with ALS within 36 months of symptom onset.
* Subjects must be ambulatory (i.e., must not be confined to a wheelchair).
* Capable of giving signed informed consent.
* Capable and willing to comply with the requirements of the protocol (either by themselves or with assistance).

Exclusion Criteria:

* The study will recruit individuals with a recent diagnosis of ALS.

Inclusion criteria:

* Aged 18 years of age or above at the time of signing the informed consent.
* Diagnosed with ALS by a neurologist with expertise in ALS (Brooks et al., 2000). For subjects with bulbar onset there must be objective limb involvement of at least one limb.
* Diagnosed with ALS within 36 months of symptom onset.
* Subjects must be ambulatory (i.e., must not be confined to a wheelchair).
* Capable of giving signed informed consent.
* Capable and willing to comply with the requirements of the protocol (either by themselves or with assistance).

Exclusion criteria:

* Neurological (other than the subject's ALS) or non-neurological co-morbidities (e.g., joint disease, respiratory disease) which limit mobility.
* Clinically significant cognitive impairment in the opinion of the investigator or lacking capacity in accordance with the Mental Capacity Act (2005).
* Regionally restricted forms of ALS, or other atypical variants:
* Isolated corticobulbar pattern of ALS with normal ambulation
* Primary lateral sclerosis
* Signs of chronic partial denervation restricted to a single limb
* ALS or parkinsonism dementia complex
* Subjects requiring mechanical ventilation (non-invasive ventilation for sleep apnoea is allowed).
* Historical or current evidence of clinically significant uncontrolled disease which, in the opinion of the chief investigator, would put the safety of the subject at risk through participation or impact the study assessments or endpoints.
* Presence of an active implantable cardiac medical device (e.g., pacemaker or implantable cardioverter-defibrillator) or at a high risk for needing external defibrillation.
* History of skin hypersensitivity to adhesives.
* Current participation in a clinical trial which in the opinion of the chief investigator might impact the objectives of this study.
* Does not have Wifi/stable internet in the home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of amyotrophic lateral sclerosis recruited through King's College Hospital's Motor Nerve Clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
EMG activity | 1 year
  Number of fasciculations from electromyography

SECONDARY OUTCOMES:
Nocturnal Respiration | 1 year
  Respiratory rate recorded from an under mattress sensor
Nocturnal heart rate | 1 year
  Heart rate recorded from an under mattress sensor
Household movement | 1 year
  Movement within the home collected from passive infrared sensors
Sleep stage ratios | 1 year
  Awake periods, light sleep, deep sleep and rapid eye movement sleep recorded from an under mattress sensor.
Blood pressure | 1 year
  Blood pressure recorded from a wireless internet enabled blood pressure monitor
Blood oxygen saturation | 1 year
  Blood oxygen saturation recorded from a smart watch
Heart beat irregularity | 1 year
  R wave cycle count from electrocardiogram within smart watch
Temperature | 1 year
  Recorded from an internet enabled thermometer
Weight | 1 year
  Recorded from smart scales
Step count | 1 year
  Step count recorded from a smart watch

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: KCL SPIQE group information — http://www.kcl.ac.uk/spiqe
- See also: Minder remote monitoring platform — https://mindermeetingplace.com/